CLINICAL TRIAL: NCT01756586
Title: Dexamethasone and Lower Extremity Block Duration
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no logistical support to carry out the study fairly
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB12-2198
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Analgesia Duration
Keywords: popliteal block; analgesia duration
MeSH Terms: interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Plain bupivacaine
  Interventions: Drug: Bupivacaine
- Experimental (Experimental): Bupivacaine with Dexamethasone
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Experimental
Drug: Bupivacaine — Control

SUMMARY:
Dexamethasone has shown to prolong upper extremity blocks. No one ha studied its effect on lower extremity blocks. The study would evaluate that point.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. foot surgery
3. no contraindication to regional anesthesia

Exclusion Criteria:

1. opioid dependent
2. chronic pain condition
3. peripheral neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Bupivacaine with Dexamethasone
  Dexamethasone
  Bupivacaine: Control
Period: Overall Study
Arm/Group | Control | Experimental
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Increase in the Duration of Block
Time Frame: 3 days
Population: Did not have resources to follow up with the subjects after the surgery. The study was terminated early.
Arm/Group | Control | Experimental
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No